CLINICAL TRIAL: NCT02531204
Title: Pharmacodynamic Study of ASP1585 - Verification of Bioequivalence Between ASP1585 Granules and ASP1585 Capsules
Brief Title: A Study of ASP1585 to Evaluate the Bioequivalence Between ASP1585 Granules and ASP1585 Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1585-CL-0201
Record Dates: First submitted 2015-08-12; First posted 2015-08-24 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Healthy; Urine Phosphorus Excretion
Keywords: ASP1585; Bioequivalence; Pharmacodynamic; Phosphate binder; Bixalomer; urinary phosphorus excretion
MeSH Terms: interventions — bixalomer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP1585 granules preceding group (Experimental)
  Interventions: Drug: ASP1585
- ASP1585 capsules preceding group (Active Comparator)
  Interventions: Drug: ASP1585

INTERVENTIONS:
Drug: ASP1585 — oral
  Other Names: Bixalomer; Kiklin

SUMMARY:
The purpose of this study is to assess the bioequivalence between ASP1585 granules and ASP1585 capsules after repeated oral administration of ASP1585 granules or ASP1585 capsules under open-label conditions in non-elderly healthy male subjects. In addition, the safety of these products is assessed.

ELIGIBILITY:
Inclusion Criteria:

* Body weight (at screening) ≥ 50.0 kg and < 80.0 kg
* Body mass index (BMI) (at screening) ≥ 17.6 kg/m2 and < 26.4 kg/m2
* Healthy, as judged by the investigator/sub-investigator based on medical history and the results of physical examination (subjective symptoms and objective findings) and all tests obtained at screening and during the period from hospital admission to immediately before study medication in 1st period.

Exclusion Criteria:

* Received or scheduled to receive any investigational drugs in other clinical trials, post-marketing studies, or clinical studies within 120 days before the screening or during the period from the screening to 1st hospitalization.
* Donated or scheduled to donate 400 mL of whole blood within 90 days before the screening or during the period from the screening to 1st hospitalization, 200 mL of whole blood within 30 days before the screening or during the period from the screening to 1st hospitalization, or blood components within 14 days before the screening or during the period from the screening to 1st hospitalization.
* Any deviation of the laboratory tests at screening or 1st hospitalization.
* A deviation from the normal range of blood pressure, pulse rate, or body temperature at screening or 1st hospitalization

  * Sitting blood pressure: Systolic blood pressure: ≥90 mmHg, ≤140 mmHg; Diastolic blood pressure: ≥40 mmHg, ≤90 mmHg
  * Sitting pulse rate; ≥40 bpm, ≤99 bpm
  * Axillary body temperature; ≥35.0°C, ≤37.0°C
* History of drug allergies
* Upper gastrointestinal disease (e.g., nausea, vomiting, and stomachache) within 7 days before 1st hospitalization
* Concurrent or previous hepatic disease (e.g., viral hepatitis, drug-induced liver injury, and hepatic impairment)
* Concurrent or previous heart disease (e.g., congestive heart failure, angina pectoris, and arrhythmia requiring treatment)
* Concurrent or previous GI disease (e.g., ileus paralytic, gastric atony, intestinal atony, colitis ulcerative, peptic ulcer and gastroesophageal reflux esophagitis; except for a history of appendicitis).
* Concurrent or previous renal disease (e.g., acute renal failure, glomerulonephritis, and interstitial nephritis)
* Concurrent or previous renal disease (e.g., acute renal failure, glomerulonephritis, and interstitial nephritis)
* Concurrent or previous cerebrovascular disorder (e.g., cerebral infarction)
* Previous use of bixalomer
* Excessive smoking or drinking habit

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Average daily amount of urine phosphorus change from baseline | Day 5 to Day 8 after start of each dosing
  Average daily amount of urine phosphorus on Day 5 to Day 8 was compared with that on Day -4 to Day 1 (baseline)

SECONDARY OUTCOMES:
Safety profile assessed by the incidence of adverse events, vital signs, clinical laboratory tests, and 12-lead ECG | Up to Day 17 on Period 2
  ECG: Electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Kagoshima, Japan